CLINICAL TRIAL: NCT02111590
Title: The Influence of Immunoglobulin Dosage and Administration on Development of Hemolytic Anemia and Variation on Muscle Strength in Patients With CIDP and MMN
Brief Title: Immunoglobulin Dosage and Administration Form in CIDP and MMN
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Octapharma Pharmazeutika Produktionsges.m.b.H. (Unknown)
Responsible Party: Principal Investigator, Johannes Jakobsen, Professor, Rigshospitalet, Denmark
Other Study IDs: 2013-400-RH
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Multifocal Motor Neuropathy; Hemolytic Anemia
Keywords: Immunoglobulins, Intravenous; Immunoglobulins, Subcutaneous
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Anemia, Hemolytic | interventions — Immunoglobulins; Injections, Subcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IVIG to SCIG: Patients with CIDP or MMN in maintenance therapy with IVIG every 3rd to 6th week are shifted to weekly SCIG treatment in unaltered dose.
  Interventions: Drug: Immunoglobulins
- SCIG to SCIG: Patients with CIDP or MMN in maintenance therapy with SCIG (Subcuvia(R) or Hizentra(R)) are shifted to treatment with Gammanorm(R) in unaltered weekly dose.
  Interventions: Drug: Immunoglobulins

INTERVENTIONS:
Drug: Immunoglobulins — SCIG dosage is individualized for each patient according to previous IVIG dosage
  Other Names: Gammanorm(R), immunoglobulin for subcutaneous use

SUMMARY:
The aim of this study is to evaluate development of hemolysis and the variation in isokinetic muscle strength in two groups of patients with chronic inflammatory demyelinating polyneuropathy (CIDP) or multifocal motor neuropathy (MMN)

1. Patients shifted from 3- or 6-weekly treatment with intravenous immunoglobulin (IVIG) to weekly treatment with subcutanoeus immunoglobulin (SCIG)
2. Patients shifted from SCIG treatment with Subcuvia® or Hizentra® to Gammanorm®.

Hypotheses

* During treatment with IVIG blood hemoglobin will fluctuate with a decline due to infusion, whereas it will remain stable during SCIG treatment without fluctuation
* Isokinetic muscle strength in affected muscle groups is more stable during treatment with SCIG than with IVIG
* Blood hemoglobin and changes in muscle strength is comparable during Subcuvia® or Hizentra® and Gammanorm® treatment

DETAILED DESCRIPTION:
Due to planned switch of treatment with immunoglobulin at Department of neurology (Rigshospitalet) patients treated with IVIG will be shifted to treatment with SCIG with an unaltered dosage. The medication is administered at home two or three times weekly. IVIG is often administered every 3 to 6 weeks. All patients will be trained in managing the treatment with SCIG by a nurse from the neurological department. When the patient is able to manage the treatment regimen it can be done at home.

All patients will be evaluated eight times during the study period. Four times before and four times after shift of treatment.

Prior to participation the intervals will be standardized to 3 or 6 weeks giving an extra infusion for those with an interval of 3 weeks, i.e. patients on 4-week interval will be switched to 3-week interval while patients on 5-week interval will be switched to 6-week interval. The dose will be adjusted leading to an unchanged weekly dose of IVIG. All patients will be evaluated in connection to two IVIG infusions. For those receiving 3 infusions examinations will be executed before and 2 weeks after the first and last infusion. SCIG is initiated 2 weeks after the last IVIG infusion.

Patients on maintenance therapy with Subcuvia® or Hizentra® will be shifted to treatment with Gammanorm® according to guidelines from the Danish Healthcare Society, the weekly dose of immunoglobulin being unaltered. They will be evaluated 3 times (once before, at the time of shift of SCIG and once after).

All evaluations at each time point in both groups consist of measurement of isokinetic muscle strength of four affected muscle groups and blood sampling detecting blood hemoglobin and hemolytic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CIDP or MMN fulfilling the EFNS/PNS criteria
* Maintenance treatment with IVIG or SCIG for at least 3 months
* Negative result on a pregnancy test (HCG-based assay in urine) for women of childbearing potential and use of a reliable method of contraception for the duration of the study

Exclusion Criteria:

* Pure sensory or severe ataxic CIDP
* Other cause of neuropathy (incl. pressure neuropathy)
* Known history of adverse reactions to IgA in other products
* Exposure to blood or any blood product or plasma derivatives, other than Privigen, within the past 3 months prior to first infusion of Gammanorm
* Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products.
* Requirement of any routine premedication for IgG administration
* History of malignancies of lymphoid cells and immunodeficiency with lymphoma
* Severe liver function impairment (ALAT 3 times above upper limit of normal)
* Known protein-losing enteropathies or proteinuria.
* Live viral vaccination (such as measles, rubella, mumps and varicella) within the last 2 months prior to first infusion of Gammanorm
* Treatment with any investigational medicinal product within 3 months prior to first infusion of Gammanorm
* Medication interfering with hematopoiesis
* Other immunomodulation therapy than low dose steroid (Prednisolone < 25 mg daily)
* Known or suspected to abuse alcohol, drugs, psychotropic agents or other chemicals within the past 12 months prior to first infusion of Gammanorm
* Known or suspected HIV, HCV, or HBV infection
* Pregnant or nursing women
* Planned pregnancy during course of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CIDP or MMN in maintenance treatment with immunoglobulins
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Variation in blood hemoglobin during treatment with IVIG and SCIG | Twenty weeks
  Patients in treated with IVIG every 6th week are shifted to weekly SCIG treatment in unaltered dose. Blood hemoglobin is measured according to two IVIG infusions, before and two weeks after, and four times with the same intervals during SCIG treatment. SCIG treatment is initiated in week 8.
  Blood samples are collected at the following time points:
  Week 0, 2, 6, 8, 12, 14, 18 and 20

SECONDARY OUTCOMES:
Variation in muscle strength during treatment with two preparations of SCIG | Twenty weeks
  Patients treated with SCIG (Subcuvia(R) or Hizentra(R)) are shifted to treatment with Gammanorm(R) in unaltered weekly dose. Muscle strength are evaluated at enrolment and after 10 weeks of treatment with (Subcuvia(R) or Hizentra(R)) and after 10 weeks of treatment with Gammanorm(R). Treatment is shifted in week 10.
  Muscle strength is meaured at the following time points:
  Week 0, 10 and 20
Variation in muscle strength during treatment with IVIG and SCIG | Twenty weeks
  Patients in treated with IVIG every 6th week are shifted to weekly SCIG treatment in unaltered dose. Isokinetic muscle strength is measured according to two IVIG infusions, before and two weeks after, and four times with the same intervals during SCIG treatment. SCIG treatment is initiated in week 8.
  Muscle strength is measured at the following time points:
  Week 0, 2, 6, 8, 12, 14, 18 and 20
Variation in blood hemoglobin during treatment with two preparations of SCIG | Twenty weeks
  Patients treated with SCIG (Subcuvia(R) or Hizentra(R)) are shifted to treatment with Gammanorm(R) in unaltered weekly dose. Blood hemoglobin is measured at enrolment and after 10 weeks of treatment with (Subcuvia(R) or Hizentra(R)) and after 10 weeks of treatment with Gammanorm(R). Treatment is shifted in week 10.
  Blood samples are collected at the following time points:
  Week 0, 10 and 20

OTHER OUTCOMES:
Comparison of Quality of life | Twenty weeks
  1. Patients in treated with IVIG every 6th week are shifted to weekly SCIG treatment in unaltered dose. Quality of life is measured by SF-36 questionaire. SCIG treatment is initiated in week 8.
     SF-36 is handed out at the following time points:
     Week 0, 8 and 20
  2. Patients treated with SCIG (Subcuvia(R) or Hizentra(R)) are shifted to treatment with Gammanorm(R) in unaltered weekly dose. Quality of life is measured by SF-36 questionaire. Treatment regimen is shifted in week 10.
  SF-36 is handed out at the following time points:
  Week 0, 10 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Jakobsen, DMSc, Principal Investigator — Neuroscience Center, Rigshospitalet
Locations (1):
- Department of Neurology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Christiansen I, Markvardsen LH, Jakobsen J. Comparisons in fluctuation of muscle strength and function in patients with immune-mediated neuropathy treated with intravenous versus subcutaneous immunoglobulin. Muscle Nerve. 2018 Apr;57(4):610-614. doi: 10.1002/mus.25967. Epub 2017 Nov 18. PMID 28881389